CLINICAL TRIAL: NCT01471561
Title: Retrospective Analysis of Cataract Surgery-induced Dry Eye Using Tear Osmolarity Testing
Brief Title: Analysis of Cataract Surgery Induced Dry Eye
Status: Completed | Type: Observational
Sponsor: TearLab Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TP00099
Record Dates: First submitted 2011-11-10; First posted 2011-11-16 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Cataract
Keywords: Osmolarity; Cataract; Dry Eye
MeSH Terms: conditions — Cataract; Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective study to determine if rates of osmolarity and dry eye disease symptoms increase following cataract surgery.

DETAILED DESCRIPTION:
The objective of this study is to determine if tear osmolarity is a good predictor for dry eye following cataract surgery.

The practice will retrospectively identify patients that have had cataract surgery from billing records. This will be cross referenced with patients that have had the diagnosis of dry eye and have had tear osmolarity testing, also from billing or electronic records analysis. The studies will be done at sites that have inclusion of a general statement about record review for research in the patient intake information at the practice. Information will be taken from the baseline visit at the final pre-operative examination prior to cataract surgery from these patients who have had tear osmolarity measured on each eye using the TearLab osmolarity device.

Because this is a retrospective study, patients will have followed each surgeon's typical pre-operative and post-operative protocol (i.e., lid cleansing, topical antibiotics, steroids, NSAIDS, etc.) without other peri-surgical complications, and followed at the normal post-operative follow-up appointments. Whenever tear osmolarity measurements had been taken and recorded in the patient's chart, this information will be collected from the patient's chart and recorded in a database. Information from visits up to and including the 3 month postoperative interval will be recorded. Additional information recorded will be demographic information such as age, corrected vision before and after the cataract surgery at the one month visit as well as at any time that tear osmolarity is measured. Additionally, any comments made in the history of present illness statement regarding dryness will be recorded in the database. Presence of other ocular surface disease present such as blepharitis, allergic disease, or anterior basement membrane dystrophy will be recorded. Systemic medications that the patient is taking will also be recorded. Presence or absence of diabetes mellitus will also be recorded. The database will be kept in a password protected computer in a locked office location, and every precaution will be taken to prevent identification of any patient specific identifiers. Information will be de-identified as soon as possible by using codes to identify the data rather than patient names or chart numbers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, eighteen years of age or older
2. Confirmed diagnosis of cataract with cataract surgery performed in at least one eye

Exclusion Criteria:

1. Any complications of cataract surgery that have required a sclera incision rather than a clear corneal incision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Male or female, eighteen years of age or older
  2. Confirmed diagnosis of cataract with cataract surgery performed in at least one eye
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Post surgical tear osmolarity | 90-Day post-surgical
  Correlation between pre-surgery value and development of dry eye disease post surgery
  1) Comparison of Osmolarity measurement pre to post-op, as well as over time, to determine change and statistical significance

SECONDARY OUTCOMES:
Post-surgical dry eye symptoms | 90-Day post-surgical
  Correlation between pre-surgery value and development of dry eye disease post surgery.
  1) Subjective patient reporting on dry eye symptoms from pre to postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Gaston Lacayo, MD, Principal Investigator
Locations (4):
- United States (4):
  - William Trattler, MD, Miami, Florida
  - David Hardten, MD, Minneapolis, Minnesota
  - Chris Starr, MD, New York, New York
  - Eric Donnenfeld, MD, Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: No
No data will be shared.